CLINICAL TRIAL: NCT02662231
Title: Determining the Worldwide Epidemiology of Surgical Site Infections After Gastrointestinal Surgery
Acronym: GlobalSurg 2
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: University of Birmingham (Other)
Responsible Party: Sponsor
Other Study IDs: GlobalSurg 2 Edinburgh
Record Dates: First submitted 2016-01-05; First posted 2016-01-25 (Estimated); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Surgical Wound Infection
Keywords: Surgical Site Infection; General Surgery; Laparotomy; Outcome and Process Assessment (Health Care); Developing Countries; International Cooperation; Specialties, Surgical; Developed Countries; Quality of Health Care
MeSH Terms: conditions — Surgical Wound Infection | interventions — Emergency Service, Hospital

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Emergency, or elective gastrointestinal resection — Gastrointestinal resection is defined as complete transection and removal of a segment of the oesophagus, stomach, small bowel, colon or rectum, including cholecystectomy, and appendicectomy.

SUMMARY:
Surgical site infection (SSI) is the most common complication following major gastrointestinal surgery, affecting between 25-40% of patients. The rate of SSI doubles from low-income to high-income settings, persisting after risk adjustment. Investigating the diagnosis and treatment of SSIs remains a largely unaddressed global health priority. The impact of antibiotic resistant organisms and the effectiveness of antibiotic prophylaxis are unknown. This study aims to determine SSI rates following gastrointestinal surgery across worldwide hospital settings.

DETAILED DESCRIPTION:
The burden of surgically disease in low and middle-income countries (LMICs) is growing. Specific programmes have aimed to raise the profile of safe surgery and anaesthesia on the global health agenda. The Lancet Commission on Global Surgery have outlined six core indicators for the assessment of global surgical systems, including the postoperative mortality rate (POMR). Although mortality is the most extreme outcome of surgery, it only affects 1-4% of all patients. For major gastrointestinal surgery, efforts to quantify POMR alone neglect the associated morbidity, which is likely to affect a far greater proportion of patients [1]. More relevant markers of postoperative outcome are needed for the majority of patients, who will survive surgery.

Surgical site infection (SSI) is the most common complication following major gastrointestinal surgery, affecting between 25-40% of patients after midline laparotomy in high-income settings, and affects both adults and children. The effects of SSI can be life threatening. They are related to one-third of postoperative deaths and accounts for 8% of all deaths caused by a nosocomial infection. Furthermore, SSIs cause pain and discomfort, increasing the time taken to return home thus further amplifying the patient's potential nosocomial infection risk. This has an important economic impact. In the UK, hospital length of stay is doubled, with an attributable cost of £30 million per year.

The 2014 prospective, observational cohort study (GlobalSurg-1) included 10,475 patients from 58 countries. It showed that the incidence of SSI more than doubled from high (7.4%), to middle (14.4%), to low (20.0%) income countries. This persisted after multivariable risk adjustment for patient and hospital confounders (middle income: odds ratio 1.96 [1.63-2.32] and low income: 2.06 [1.67-2.57]). In the most contaminated and dirty operations, one in three patients from LMICs suffered an SSI. Dirty surgery doubled in low-income countries (29.7% versus 16.6% in high-income settings), which was in turn associated with doubling of SSI (34.5% low-income versus 15.4% high-income). However, SSI was assessed as a secondary outcome measure as part of that study, lacking validity and requiring external validation.

Antibiotic resistant organisms are now prevalent worldwide and a focus of interest for policy leaders and global health advocates. Some hospitals have no information on the rate of antibiotic resistant SSIs. For those patients who contract infections caused by resistant organisms, they are posed with a higher risk of mortality, morbidity and require more healthcare resources. Currently no data exists to describe the international epidemiology of SSIs, their causative organisms and drug-resistance. Therefore, investigating the diagnosis and treatment of SSIs is an urgent global health priority.

The primary aim of this study is to determine SSI rates across low, middle and high Human Development Index (HDI) countries. The secondary aims include describing organisms causing SSI rates, use of microbiologic tests, and rate of antibiotic resistant SSI. The impact of the method of 30-day follow-up on these outcomes will also be analysed. Other aims include describing the burden of surgical disease using 30-day mortality rates, perforated appendicitis rates and laparoscopic cholecystectomy rates.

ELIGIBILITY:
Centre Inclusion Criteria:

* Any surgical unit worldwide is eligible to enter
* All participating centres will be required to register their details, complete an online training module, and complete a pilot audit prior to commencing
* Centres must ensure that they can include consecutive patients and provide at least 95% data completeness
* There is no minimum number of patients per centre, as long as the patient(s) included are consecutive

Inclusion criteria:

* Patients of all ages (adult and paediatric)
* Consecutive patients during a chosen 14-day study period
* Undergoing emergency or elective gastrointestinal resection, cholecystectomy and appendectomy.
* Includes open, laparoscopic, laparoscopic converted and robotic cases
* Primary indication of trauma should be included
* Hernia repair with bowel resection should be included

Exclusion criteria:

* Operations with a primary indication that is vascular, gynaecological, urological (including ileal conduit) or transplant
* Caesarean sections
* Whipples procedure
* Simple hernia repair

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive patients undergoing emergency, or elective gastrointestinal resection, cholecystectomy and appendectomy.
Sampling Method: Probability Sample
Enrollment: 12539 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-07-31 (Actual); Study Completion 2016-09-30 (Actual)

PRIMARY OUTCOMES:
Superficial incisional surgical site infection (SSI) | Within 30 days of surgery
  This measure adapts the definitions within the 2008 Centre for Disease Control definitions of SSI.

SECONDARY OUTCOMES:
Postoperative mortality rate (POMR) | Within 30 days of surgery
  Death any time after skin incision until the 30th day after surgery. If the patient is discharged alive but not seen again by day 30, this is equivalent to the in-patient mortality rate.
Postoperative re-intervention rate | Within 30 days of surgery
  Operative, radiological or endoscopic re-intervention any time after skin incision until the 30th day after surgery. If the patient is discharged alive but not seen again by day 30, this is equivalent to the inpatient re-intervention rate.
Rate of antibiotic-resistant surgical site infection | Within 30 days of surgery
  Describing international variation, where available.
Organism causing surgical site infection | Within 30 days of surgery
  Patient-level, online questionnaire. Organisms identified upon microscopy and culture. Grouped by recognised causative bacteria in superficial surgical site infection (i.e. Staphylococcus Aureus, Coliform, Anaerobe, Other)
Proportion of patients treated in a hospital with microscopy, culture and sensitivity testing | Within 30 days of surgery
  Patient-level, online questionnaire.

OTHER OUTCOMES:
Follow up method for detecting surgical site infection | Within 30 days of surgery
  Assessing method used to detect SSI at thirty day review (i.e. still an inpatient, clinic review, telephone review, community/home review, discharged before 30 days and not contacted again)
Complicated appendicitis rate | Pre-, or intra-operatively
  Includes radiological or clinical perforation of the appendix, empyema or abscess formation, and fecal peritonitis.
Laparoscopic cholecystectomy rate | Intra-operatively

CONTACTS AND LOCATIONS:
Overall Officials: Aneel Bhangu, Principal Investigator — University of Birmingham; Ewen M Harrison, Principal Investigator — University of Edinburgh; Edward Fitzgerald, Principal Investigator — Royal Free London NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Royal Infirmary of Edinburgh, Edinburgh

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be made available upon request, to enable patient level meta-analysis

REFERENCES:
- [Background] Pearse RM, Moreno RP, Bauer P, Pelosi P, Metnitz P, Spies C, Vallet B, Vincent JL, Hoeft A, Rhodes A; European Surgical Outcomes Study (EuSOS) group for the Trials groups of the European Society of Intensive Care Medicine and the European Society of Anaesthesiology. Mortality after surgery in Europe: a 7 day cohort study. Lancet. 2012 Sep 22;380(9847):1059-65. doi: 10.1016/S0140-6736(12)61148-9. PMID 22998715
- [Background] Bhangu A, Fitzgerald JE, Fergusson S, Khatri C, Holmer H, Soreide K, Harrison EM. Determining universal processes related to best outcome in emergency abdominal surgery: a multicentre, international, prospective cohort study. BMJ Open. 2014 Oct 29;4(10):e006239. doi: 10.1136/bmjopen-2014-006239. PMID 25354824
- [Background] Pinkney TD, Calvert M, Bartlett DC, Gheorghe A, Redman V, Dowswell G, Hawkins W, Mak T, Youssef H, Richardson C, Hornby S, Magill L, Haslop R, Wilson S, Morton D; West Midlands Research Collaborative; ROSSINI Trial Investigators. Impact of wound edge protection devices on surgical site infection after laparotomy: multicentre randomised controlled trial (ROSSINI Trial). BMJ. 2013 Jul 31;347:f4305. doi: 10.1136/bmj.f4305. PMID 23903454
- [Background] Wilson AP, Gibbons C, Reeves BC, Hodgson B, Liu M, Plummer D, Krukowski ZH, Bruce J, Wilson J, Pearson A. Surgical wound infection as a performance indicator: agreement of common definitions of wound infection in 4773 patients. BMJ. 2004 Sep 25;329(7468):720. doi: 10.1136/bmj.38232.646227.DE. Epub 2004 Sep 14. PMID 15367425
- [Background] Horan TC, Andrus M, Dudeck MA. CDC/NHSN surveillance definition of health care-associated infection and criteria for specific types of infections in the acute care setting. Am J Infect Control. 2008 Jun;36(5):309-32. doi: 10.1016/j.ajic.2008.03.002. No abstract available. PMID 18538699
- [Background] Laxminarayan R, Duse A, Wattal C, Zaidi AK, Wertheim HF, Sumpradit N, Vlieghe E, Hara GL, Gould IM, Goossens H, Greko C, So AD, Bigdeli M, Tomson G, Woodhouse W, Ombaka E, Peralta AQ, Qamar FN, Mir F, Kariuki S, Bhutta ZA, Coates A, Bergstrom R, Wright GD, Brown ED, Cars O. Antibiotic resistance-the need for global solutions. Lancet Infect Dis. 2013 Dec;13(12):1057-98. doi: 10.1016/S1473-3099(13)70318-9. Epub 2013 Nov 17. PMID 24252483
- [Background] Earnshaw S, Mendez A, Monnet DL, Hicks L, Cruickshank M, Weekes L, Njoo H, Ross S. Global collaboration to encourage prudent antibiotic use. Lancet Infect Dis. 2013 Dec;13(12):1003-4. doi: 10.1016/S1473-3099(13)70315-3. Epub 2013 Nov 17. No abstract available. PMID 24252477
- [Background] Tanner J, Khan D, Aplin C, Ball J, Thomas M, Bankart J. Post-discharge surveillance to identify colorectal surgical site infection rates and related costs. J Hosp Infect. 2009 Jul;72(3):243-50. doi: 10.1016/j.jhin.2009.03.021. Epub 2009 May 15. PMID 19446918
- [Background] Plowman R, Graves N, Griffin MA, Roberts JA, Swan AV, Cookson B, Taylor L. The rate and cost of hospital-acquired infections occurring in patients admitted to selected specialties of a district general hospital in England and the national burden imposed. J Hosp Infect. 2001 Mar;47(3):198-209. doi: 10.1053/jhin.2000.0881. PMID 11247680
- [Background] Coello R, Charlett A, Wilson J, Ward V, Pearson A, Borriello P. Adverse impact of surgical site infections in English hospitals. J Hosp Infect. 2005 Jun;60(2):93-103. doi: 10.1016/j.jhin.2004.10.019. PMID 15866006
- [Background] Smyth ET, McIlvenny G, Enstone JE, Emmerson AM, Humphreys H, Fitzpatrick F, Davies E, Newcombe RG, Spencer RC; Hospital Infection Society Prevalence Survey Steering Group. Four country healthcare associated infection prevalence survey 2006: overview of the results. J Hosp Infect. 2008 Jul;69(3):230-48. doi: 10.1016/j.jhin.2008.04.020. Epub 2008 Jun 11. PMID 18550218
- [Background] Meara JG, Greenberg SL. The Lancet Commission on Global Surgery Global surgery 2030: Evidence and solutions for achieving health, welfare and economic development. Surgery. 2015 May;157(5):834-5. doi: 10.1016/j.surg.2015.02.009. No abstract available. PMID 25934019
- [Derived] NIHR Global Health Research Unit on Global Surgery, GlobalSurg Collaborative. Use of Telemedicine for Postdischarge Assessment of the Surgical Wound: International Cohort Study, and Systematic Review With Meta-analysis. Ann Surg. 2023 Jun 1;277(6):e1331-e1347. doi: 10.1097/SLA.0000000000005506. Epub 2022 Jun 27. PMID 36626409
- [Derived] GlobalSurg Collaborative. Surgical site infection after gastrointestinal surgery in high-income, middle-income, and low-income countries: a prospective, international, multicentre cohort study. Lancet Infect Dis. 2018 May;18(5):516-525. doi: 10.1016/S1473-3099(18)30101-4. Epub 2018 Feb 13. PMID 29452941
- [Derived] GlobalSurg Collaborative. Determining the worldwide epidemiology of surgical site infections after gastrointestinal resection surgery: protocol for a multicentre, international, prospective cohort study (GlobalSurg 2). BMJ Open. 2017 Jul 21;7(7):e012150. doi: 10.1136/bmjopen-2016-012150. PMID 28733294
- See also: GlobalSurg-II Project Hub — http://globalsurg.org/projects/globalsurg-2/
- Available data/document: Study Protocol — http://globalsurg.org/globalsurg-2-protocol/ — GlobalSurg-II Study Protocol: available in multiple languages